CLINICAL TRIAL: NCT06410430
Title: Exploration the Therapeutic Mechanism of Ba-Duan-Jin in the Treatment of Fibromyalgia by Improving Gut Microbiota and Brain Magnetic Resonance Imaging
Brief Title: Exploration the Mechanism of Ba-Duan-Jin in the Treatment of Fibromyalgia Based on Brain-gut Axis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Juan Jiao, Chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CI2021A0151
Record Dates: First submitted 2024-04-24; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ba-Duan-Jin group (Experimental): The participants will be trained and guided online by an experienced Ba-Duan-Jin instructor with reference to the standard operating procedure (SOP) for a 12-week course of 1 hour twice a week.
  Interventions: Behavioral: Ba-Duan-Jin
- Healthy control group (No Intervention)

INTERVENTIONS:
Behavioral: Ba-Duan-Jin — Ba-Duan-Jin is a common form of "self-healthcare" Qigong exercise that has been practiced by Chinese people for at least eight hundred years.It consists of eight sets of simple movements. By combining meditation with slow, graceful ovements,deep breathing, and relaxation, Ba-Duan-Jin practitioners believe it has the ability to move vital energy (Qi) throughout the body. Ba-Duan-Jin is also considered to be a multicomponent intervention that integrates physical, psychosocial, emotional, spiritual, and behavioral elements. While the biological mechanisms remain unclear.
  Other Names: Baduanjin; Eight Brocades; Eight-Section Brocade
  Arms: Ba-Duan-Jin group

SUMMARY:
To investigate the mechanism by Ba-Duan-Jin in the treatment of fibromyalgia. Twenty eligible fibromyalgia patients were selected, and were trained and guided online by an experienced Ba-Duan-Jin instructor with reference to the standard operating procedure (SOP) for a 12-week course of 1 hour twice a week. The evaluation points were 0, 4, 8, and 12 weeks. The change of pain Visual Analogue Score (VAS) and tener point count (TPC) post-treatment were evaluated. And blood, feces, and brain fMRI were collected from the patients at 0 and 12 weeks to compare the changes in gut microbiota, metabolites, and brain function networks before and after the intervention with the 16SrRNA sequencing, targeted metabolomics, and real-time Quantitative Polymerase Chain Reaction (PCR).

ELIGIBILITY:
Inclusion Criteria:

* Meet the 1990 American College of Rheumatology (ACR) Research Classification Criteria for fibromyalgia or 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria;
* Be over 18 years of age;
* Female;
* Right-handedness;
* Sign informed consent.

Exclusion Criteria:

* be less than 40mm of pain VAS score;
* had received any treatments for fibromyalgia or probiotic bacteria within 2 weeks;
* had received antibiotics within 4 weeks;
* had practiced Ba-Duan-Jin, Tai Chi, yoga, or other forms of Qigong within previous 12 months;
* had severe depression or anxiety;
* pregnancy or planned pregnancy within the study period;
* had any poorly-controlled comorbid medical conditions, such as dementia, cancer, thyroid disease, inflammatory arthritis;
* patients with a history of head trauma, cerebral infarction or cerebral haemorrhage
* contraindications for MRI,including metal implants, cardiac pacemaker,false tooth, surgical artery clips, metal tattoos or claustrophobia;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The change of the Visual Analogue Scale (VAS) for pain from baseline | Baseline, week4, week8, week12
  Pain VAS, range from 0 to 100 mm with higher score indicating more severe pain
The change of Tender Point Count (TPC) from baseline | Baseline, week4, week8, week12
  TPC, the 18 body points of the 1990 American College of Rheumatology (ACR) Research Classification Criteria for fibromyalgia, which in healthy subjects do not cause pain, whereas in patients with fibromyalgia no fewer than 11 are painful

SECONDARY OUTCOMES:
Gut microbiota sequencing results by analyzing metagenomes of microbial genes | Baseline, week12
  Fecal samples are obtained from the Ba-Duan-Jin group and control group. After extracting DNA from fecal samoles, high-throughput Illumina sequencing, gene classification, abundance calculation, functional and metabolic annotation will be performed on the extracted DNA. The Bowtie2, BWA and Soap2 will be selected for the comparison software.
  The condition of comparison is to obtain the comparison results of 95% identity (and above).
Serum fatty acids metabolism results by UPLC-MS/MS | Baseline, week12
  Blood samples are obtained from the Ba-Duan-Jin group and control group. Ultra Performance Liquid Chromatography Tandem Mass Spectrometry will be performed. The SIMCA will be selected for Orthogonal Partial Least Squares-Discriminant Analysis. The Kyoto encyclopedia of genes and genomes will be selected for functional enrichment analysis of differential metabolites.
Brain morphology in fibromyalgia patients measured by structural MRI | Baseline, week12
  To compare the changes in brain structure and morphology in patients with fibromyalgia before and after treatment by structural MRI. The images were acquired by a Siemens 3.0T Skyra scanner (Siemens; Munich, Germany) using fast spoiled gradient-echo sequence. Images contain whole brain, grey matter, white matter, atlas-based regions of interest for the patient group and healthy controls. The structural MRI images were processed with CAT 12 software (Version12.7, r1700). In detail, the voxel-based morphometry pipeline includes initial and refined voxel-based processing.
Brain functional connectivity in fibromyalgia patients measured by function MRI | Baseline, week12
  To compare the changes in connectivity and metabolic function of the brain in patients with fibromyalgia before and after treatment by function MRI. The scanning sequence is set up under the guidance of an imaging professional, while ensuring that the participants undergo the MRI scans with their eyes closed but awake; head movements do not exceed 1.5 mm in translation in any direction and 1.5° in rotation in any direction.
The change of the revised Fibromyalgia Impact Questionnaire (FIQR) from baseline | Baseline, week4, week8, week12
  A self-administered questionnaire with 10 subscales, measuring fibromyalgia symptoms and function domains. FIQR total score ranges from 0 to 100, with higher scores indicating more severe symptoms.
The change of the Short Form-36 Health Status Questionnaire (SF-36) from baseline | Baseline, week4, week8, week12
  The Short Form-36 Health Status Questionnaire (SF-36), which measured health-related quality of life (range, 0 to 100, with higher scores indicating better perceived health status

OTHER OUTCOMES:
The change of the Minimum Mental State Examination(MMSE) from baseline | Baseline, week4, week8, week12
  The Minimum Mental State Examination(MMSE) scores range from 0 to 30, with higher scores indicating better cognitive function
The change of the Hamilton Anxiety Scale#HAMA# from baseline | Baseline, week4, week8, week12
  The Hamilton Anxiety Scale is used to assess the severity of anxiety symptoms and consists of 14 items, with higher scores indicating greater anxiety
The change of the Multidimensional Fatigue Inventory-20 (MFI-20) from baseline | Baseline, week4, week8, week12
  The Multidimensional Fatigue Inventory-20 (MFI-20) measures fatigue severity. The MFI-20 total score ranges from 0 to 80, with higher scores indicate more severe fatigue.
The change of the Perceived Stress Scale (PSS) from baseline | Baseline, week4, week8, week12
  The Perceived Stress Scale (PSS) is for measuring the perception of stress and The Perceived Stress Scale (PSS) is for measuring the perception of stress and current levels of experienced stress. Scores range from 0 to 56, with higher total score indicating a greater degree of symptom severity
The change of the Pittsburgh Sleep Quality Index (PSQI) from baseline | Baseline, week4, week8, week12
  Scores on the Pittsburgh Sleep Quality Index (PSQI) range from 0 to 21, with higher scores indicating worse sleep quality.
The change of the Montreal Cognitive Assessment (MOCA) from baseline | Baseline, week4, week8, week12
  The MOCA scale includes visuospatial function (maximum 5 points), naming (maximum 3 points), attention ability (maximum 6points), language skills (maximum 3 points), abstract thinking ability (maximum2points), memory ability (maximum 5 points), and orientation ability (maximum 6 points), with a total score of 30 points.
The change of the Hospital anxiety and depression scale(HADS) from baseline | Baseline, week4, week8, week12
  The HADS is a 14-item, 4-point Likert scale-based self-report rating measure (with a range of 0-3). Seven questions on this scale are used to assess depression and anxiety. The sum of the 14 items determines the final score, while the specific seven items (ranging from 0 to 21) determine the final score for each subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Jiao J, Russell IJ, Wang W, Wang J, Zhao YY, Jiang Q. Ba-Duan-Jin alleviates pain and fibromyalgia-related symptoms in patients with fibromyalgia: results of a randomised controlled trial. Clin Exp Rheumatol. 2019 Nov-Dec;37(6):953-962. Epub 2019 Feb 15. PMID 30789154
- See also: Ba-Duan-Jin alleviates pain and fibromyalgia-related symptoms in patients with fibromyalgia: results of a randomised controlled trial. — http://www.clinexprheumatol.org/abstract.asp?a=13602